CLINICAL TRIAL: NCT03087305
Title: Incidence of Supraclavicular Lymph Node Metastasis in Patients Referred for EBUS-TBNA for Presumed Primary Lung Cancer by Interventional Pulmonologists.
Brief Title: Incidence of SCLN Metastasis in Patients Referred for EBUS-TBNA
Status: Withdrawn | Type: Observational
Why Stopped: low enrollment rate
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1703M10502
Record Dates: First submitted 2017-03-15; First posted 2017-03-22 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
Keywords: Interventional Pulmonary; EBUS-TBNA; Lung cancer staging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: All patients age 20yrs or greater referred for EBUS-TBNA with suspicion for primary lung cancer
  Interventions: Diagnostic Test: Supraclavicular lymph node ultrasound

INTERVENTIONS:
Diagnostic Test: Supraclavicular lymph node ultrasound — Patients will have supraclavicular lymph node assessed prior to EBUS-TBNA

SUMMARY:
Evaluation of the anatomic extent of a primary lung cancer and presence of metastasis are essential for selection of an appropriate management strategy. Endobronchial ultrasound transbronchial needle aspiration (EBUS-TBNA) is a reliable and established technique to evaluate involvement of mediastinal lymph nodes (LN); however, it is an invasive procedure and may not be tolerated in patients with severe underlying lung disease. One exception is the superficially located supraclavicular lymph nodes (SCLN), which can easily be biopsied with percutaneous US-guided-fine needle aspiration (US-FNA). Traditionally, this nodal group is evaluated by palpation; however, literature suggests that palpation itself fails to capture 66% of proven disease by cytology, which challenges the acceptance that non-palpable nodes are indicative of absent disease. Since all palpable SCLN are biopsied to rule out metastasis, we may potentially up-stage more patients using ultrasound evaluation for non-palpable nodes; and offer more appropriate management. Currently, the incidence for non-palpable SCLN metastasis has not been defined in this patient population presenting for EBUS-TBNA. The primary objective is to determine the incidence of supraclavicular lymph node metastasis by ultrasound evaluation in patients referred for EBUS-TBNA.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 20yrs or greater referred for EBUS-TBNA with suspicion for primary lung cancer

Exclusion Criteria:

1. Refusal to sign consent
2. Signs of skin infection along the neck
3. Adults who lack the capacity to sign consent.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients age 20yrs or greater referred for EBUS-TBNA with suspicion for primary lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of supraclavicular metastasis | 7 days
  Incidence of supraclavicular metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karsell PR, McDougall JC. Diagnostic tests for lung cancer. Mayo Clin Proc. 1993 Mar;68(3):288-96. doi: 10.1016/s0025-6196(12)60051-2. PMID 8474273
- [Background] Baatenburg de Jong RJ, Rongen RJ, Lameris JS, Harthoorn M, Verwoerd CD, Knegt P. Metastatic neck disease. Palpation vs ultrasound examination. Arch Otolaryngol Head Neck Surg. 1989 Jun;115(6):689-90. doi: 10.1001/archotol.1989.01860300043013. PMID 2655666
- [Background] Som PM, Curtin HD, Mancuso AA. Imaging-based nodal classification for evaluation of neck metastatic adenopathy. AJR Am J Roentgenol. 2000 Mar;174(3):837-44. doi: 10.2214/ajr.174.3.1740837. PMID 10701636
- [Background] Tsunodo-Shimizu H, Saida Y. Ultrasonographic visibility of supraclavicular lymph nodes in normal subjects. J Ultrasound Med. 1997 Jul;16(7):481-3. doi: 10.7863/jum.1997.16.7.481. PMID 9315199
- [Background] Vassallo P, Wernecke K, Roos N, Peters PE. Differentiation of benign from malignant superficial lymphadenopathy: the role of high-resolution US. Radiology. 1992 Apr;183(1):215-20. doi: 10.1148/radiology.183.1.1549675.
- [Background] Brantigan JW, Brantigan CO, Brantigan OC. Biopsy of nonpalpable scalene lymph nodes in carcinoma of the lung. Am Rev Respir Dis. 1973 Jun;107(6):962-74. doi: 10.1164/arrd.1973.107.6.962. No abstract available. PMID 4712440
- [Background] van Overhagen H, Brakel K, Heijenbrok MW, van Kasteren JH, van de Moosdijk CN, Roldaan AC, van Gils AP, Hansen BE. Metastases in supraclavicular lymph nodes in lung cancer: assessment with palpation, US, and CT. Radiology. 2004 Jul;232(1):75-80. doi: 10.1148/radiol.2321030663. Epub 2004 May 27. PMID 15166326
- [Background] Kumaran M, Benamore RE, Vaidhyanath R, Muller S, Richards CJ, Peake MD, Entwisle JJ. Ultrasound guided cytological aspiration of supraclavicular lymph nodes in patients with suspected lung cancer. Thorax. 2005 Mar;60(3):229-33. doi: 10.1136/thx.2004.029223. PMID 15741441
- [Background] Kendirlinan R, Ozkan G, Bayram M, Bakan ND, Tutar M, Gur A, Camsari G. Ultrasound guided fine-needle aspiration biopsy of metastases in nonpalpable supraclavicular lymph nodes in lung cancer patients. Multidiscip Respir Med. 2011 Aug 31;6(4):220-5. doi: 10.1186/2049-6958-6-4-220. PMID 22958429
- [Background] Chang DB, Yang PC, Yu CJ, Kuo SH, Lee YC, Luh KT. Ultrasonography and ultrasonographically guided fine-needle aspiration biopsy of impalpable cervical lymph nodes in patients with non-small cell lung cancer. Cancer. 1992 Sep 1;70(5):1111-4. doi: 10.1002/1097-0142(19920901)70:53.0.co;2-4. PMID 1325269
- [Background] Fultz PJ, Feins RH, Strang JG, Wandtke JC, Johnstone DW, Watson TJ, Gottlieb RH, Voci SL, Rubens DJ. Detection and diagnosis of nonpalpable supraclavicular lymph nodes in lung cancer at CT and US. Radiology. 2002 Jan;222(1):245-51. doi: 10.1148/radiol.2221010431. PMID 11756733
- [Background] Lee JD, Ginsberg RJ. Lung cancer staging: the value of ipsilateral scalene lymph node biopsy performed at mediastinoscopy. Ann Thorac Surg. 1996 Aug;62(2):338-41. PMID 8694587